CLINICAL TRIAL: NCT04945265
Title: Mechanistic Insight Into Ovarian Granulosa Cell Function Based on Age and Cause of Infertility
Brief Title: Effects of Age and Infertility on Ovarian Granulosa Cell Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 264510
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Infertility, Female; Infertility Unexplained; Infertility of Tubal Origin; Infertility
Keywords: ovary; granulosa cells; infertility; ageing
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Women aged <30
- Women aged 30-36
- Women aged 37-40
- Women aged >40
- Women undergoing egg freezing/male factor infertility/genetic testing
- unidentified cause of infertility
- PCOS
- endometriosis
- tubal disorders
- ovulatory disorders
- other causes of infertility e.g., fibroids.

SUMMARY:
Infertility is a life changing disorder, affecting 1 in 7 couples within the UK. Treatment options pose a significant cost burden to both the NHS and patient when NHS-funded treatment options are exhausted. This highlights the need for refinements in clinical management strategies for this patient group. Although there have been advancements in assisted reproductive technologies, the success rates of techniques such as in vitro fertilization (IVF) remain low. Surprisingly, the IVF hormonal regimens used by most assisted conception units fail to take account of patient age, ovarian reserve or cause of infertility when deciding on treatment regimen, with a 'one size fits all' approach to treatment. The investigators propose that age and cause of infertility modify the functions and environment provided by the cells (granulosa cells) that support egg (oocyte) growth and development and understanding these changes will allow for a more personalised approach to IVF treatment regimens. The aim of this study therefore is to recruit female patients undergoing IVF with different causes of infertility and age, and harvest granulosa cells from remaining material (follicular aspirates) generated at the time of egg retrieval. Granulosa cells will be cultured in vitro and cellular functions assessed. The investigators will also recruit female patients with normal fertility undergoing IVF procedure due to other reasons (i.e. egg freezing, diagnostics of genetic diseases on embryos).

ELIGIBILITY:
Inclusion Criteria:

* Any woman that is:
* fluent in English,
* capable of giving consent,
* reproductive age (between the ages of 18-45),
* is HIV and Hep A and Hep B negative.
* undergoing IVF treatment for one of the following reasons:

  1. unexplained infertility
  2. tubal disease
  3. egg freezing
  4. polycystic ovarian syndrome
  5. ovulatory disorders
  6. endometriosis
  7. male factor infertility
  8. any other cause of infertility such as fibroids.

Exclusion Criteria:

* Adults unable to consent for themselves,
* Non-fluent English speakers, unless in clinic translators are available
* Aged less than 18
* Is HIV or Hep A or B positive, or has not undergone screening.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Women undergoing routine IVF treatment as part of their clinical treatment plan.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of hormone production, protein and RNA expression | 0-14 days
  Assessed via cellular signalling responses to endocrine stimulation, production of steroid hormones, protein analysis and RNA analysis

SECONDARY OUTCOMES:
Correlation of cellular responses with age and cause of infertility. | 12 months
  Assessed via statistical analysis

IPD SHARING:
Plan to Share IPD: No